CLINICAL TRIAL: NCT00795535
Title: Heart Rate Variability in Trauma Patients
Acronym: HRV
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Kenneth Proctor, Professor, University of Miami
Other Study IDs: 20060938
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Trauma
Keywords: Injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop new triage tool for trauma patients based on HRV. EKG will be prospectively measured in trauma patients in two locations: in the prehospital setting (the field and during transport by helicopter) and in the hospital setting. In each case HRV will be derived from the EKG signal, will be correlated with other non-invasive signals (e.g. near infrared spectroscopy (NIR), and bispectral EEG (BIS)), along with other routinely measured variables (blood pressure, respiratory rate, pulse oximetry, etc), will be correlated with injury severity and day of discharge. An algorithm will be constructed using multiple linear regression. The hypotheses are:

1. reduced HRV in the field correlates with bad outcome;
2. the specificity and efficiency of HRV as a screening tool can be improved by controlling factors such as heart rate, age, gender, respiratory rate, and pulse oxygen saturation;
3. an easy to interpret HRV index can be derived that can be used for trauma triage or diagnosis.

DETAILED DESCRIPTION:
The eligible study population will be comprised of patients who meet level 1 trauma criteria and are transported by helicopter to Ryder Trauma Center or who are already admitted to the trauma center for presumptive traumatic brain injury. In addition to the EKG, trauma patients may also be connected to either an non-invasive NIR Monitor, which provides real-time information about perfusion status and/or a bispectral EEG monitor, which provides real-time information about brain metabolic activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet level 1 trauma criteria and are transported by helicopter to Ryder Trauma Center
* An additional study population will be comprised of patients already admitted to the trauma center for presumptive Traumtaic Brain Injury

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All trauma patients
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2007-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Proctor, PhD, Principal Investigator — University of Miami
Locations (1):
- Ryder Trauma Center, Miami, Florida, United States

REFERENCES:
- [Background] Proctor KG, Atapattu SA, Duncan RC. Heart rate variability index in trauma patients. J Trauma. 2007 Jul;63(1):33-43. doi: 10.1097/01.ta.0000251593.32396.df. PMID 17622866

RESULTS

PARTICIPANT FLOW:
Groups:
- Trauma Patients: Patients transported to the trauma center by helicopter
Period: Overall Study
Arm/Group | Trauma Patients
Started | 95
Completed | 75
Not Completed | 20
Not completed — incomplete data and technical problems | 20

BASELINE CHARACTERISTICS:
Population: 75 patients with complete HRV and trauma registry data
Arm/Group | Trauma Patients
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 47

OUTCOME MEASURES:

1. Primary Outcome: Base Deficit </= -6
Description: Indicator for volume deficit and resuscitation. Number of participants with Base Deficit </= -6 is reported. Base deficit is the absolute difference of the base deficit from its normal range (-2 to 2), and is used as an indicator for traumatic injuries. A base deficit </= - 6 signifies volume deficit and the need for volume resuscitation with fluids, blood or blood products either alone or in combination.
Time Frame: Upon arrival to the hospital
Population: 75 patients with complete HRV and trauma registry data
Measure: Number; unit: participants
Arm/Group | Trauma Patients
Number analyzed (Participants) | 75
participants | 12

2. Primary Outcome: Serious Injury
Description: A patient was classified as seriously injured when two of three blinded trauma surgeons classified the patient as similar after review of each patient chart and final diagnoses in retrospect.
Time Frame: Upon arrival to the hospital
Population: 75 patients with complete HRV and trauma registry data
Measure: Number; unit: participants
Arm/Group | Trauma Patients
Number analyzed (Participants) | 75
participants | 36

3. Primary Outcome: Life Saving Intervention in the Operating Room.
Description: A patient was classified as having a life saving intervention in the operating room when two of three blinded trauma surgeons classified the patient as similar after review of each patient chart and final diagnoses in retrospect.
Time Frame: Upon arrival to the hospital
Population: 75 patients with complete HRV and trauma registry data
Measure: Number; unit: participants
Arm/Group | Trauma Patients
Number analyzed (Participants) | 75
participants | 10

4. Primary Outcome: SDNN: Standard Deviation of the Normal-to-normal R-R Interval
Description: A determination of HRV derived from the time domain of a standard electrocardiogram, primarily determined by measuring the randomness of the exact occurrence of when one R wave follows a preceding R wave.
Time Frame: Upon arrival to the hospital
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Trauma Patients
Number analyzed (Participants) | 75
milliseconds (ms) | 42 (31)
Statistical Analysis 1: Comparison: Trauma Patients; Wilcoxon rank sum tests were used to compare continuous predictors, whereas chi-square tests were used to compare dichotomized predictors between those with and without serious injury. Test characteristics (specificity and positive/negative predictive values) of continuous predictors were reported based on threshold values chosen for a minimum of 80% of sensitivity. Multiple logistic regression models were used to examine the marginal effect of each predictor; Test type: Superiority or Other; p < 0.15, Wilcoxon (Mann-Whitney) — To avoid overfitting the models, only predictors with p<0.15 were included in the final models

ADVERSE EVENTS:
Time Frame: Duration of transport from injury to hospital
Arm/Group | Trauma Patients
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No